CLINICAL TRIAL: NCT00636415
Title: Intra-Articular Morphine Versus Bupivacaine on Knee Motion in Patients With Osteoarthritis: Randomized and Double-Blind Clinical Trial
Brief Title: Intra-Articular Morphine Versus Bupivacaine on Knee Motion in Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Adriana Machado Issy/ Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Intra-articular morphine; No grant
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Analgesia
Keywords: Analgesia; Morphine; Bupivacaine; Osteoarthritis; Knee
MeSH Terms: conditions — Agnosia; Osteoarthritis | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): G1 patients received morphine intra-articular route G2 patients received bupivacaine without epinephrine.
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: morphine — 1 mg (1 ml) morphine diluted in 9 ml saline by the intra-articular route, and 25 mg (10 ml) 0.25% bupivacaine without epinephrine.
  Other Names: dimorf

SUMMARY:
CONTEXT AND OBJECTIVE: Osteoarthritis causes pain and disability in a high percentage of elderly people. The aim of the present study was to compare the analgesic effect of intra-articular bupivacaine and morphine in patients with knee osteoarthritis.

DESIGN AND SETTING: A randomized and double-blind study was performed at a Pain Clinic of São Paulo Federal University.

METHODS: Thirty-nine patients with pain for more than 3 months and an intensity higher than 3 on a numerical scale (zero to 10) were included. G1 patients received 1 mg (1 ml) morphine diluted in 9 ml saline by the intra-articular route, and G2 patients received 25 mg (10 ml) 0.25% bupivacaine without epinephrine. Pain was assessed on a numerical scale and knee flexion and extension angles were measured after administration of the drugs at rest and during movement. The total amount of analgesic complementation with 500 mg paracetamol was also determined.

DETAILED DESCRIPTION:
Among the 39 patients selected, two patients from group 1 and five from group 2 were excluded from some of the analyses because they did not return on the day of assessment or because they used a complementary analgesic different from that standardized in the study

ELIGIBILITY:
Inclusion Criteria:

* Older than 50 years with a radiological confirmation of chronic knee osteoarthritis
* Pain lasting for more than 3 months either at rest or under strain, morning stiffness
* Absence of heat at the site
* Crepitation during movement and a pain score ranging from three to ten.

Exclusion Criteria:

* Patients with coagulopathy
* Infection or malignant disease
* Patients who underwent knee or hip surgery; AND
* Patients using opioids 24 hours prior to the study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2005-07 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pain relief | 1 year

SECONDARY OUTCOMES:
bupivacaine and morphine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Issy, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Pain Setor of Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gazi MB, Sakata RK, Issy AM. Intra-articular morphine versus bupivacaine for knee motion among patients with osteoarthritis: randomized double-blind clinical trial. Sao Paulo Med J. 2008 Nov;126(6):309-13. doi: 10.1590/s1516-31802008000600003. PMID 19274316